CLINICAL TRIAL: NCT01284842
Title: Call-associated Acute Fatigue in Surgical Residency- Subjective Perception or Objective Fact?
Brief Title: Call- Associated Acute Fatigue in Surgical Residency
Acronym: CAFIS
Status: Completed | Type: Observational
Sponsor: Philipps University Marburg (Other)
Responsible Party: Katja Maschuw, MD, Philipps-University Marburg, Germany
Other Study IDs: Philipps-University Marburg
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2008-06

CONDITIONS: Sleep Deprivation
Keywords: sleep-deprivation; virtual reality; residency; performance
MeSH Terms: conditions — Sleep Deprivation | interventions — CD56 Antigen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: 24-Hour-Call — one 24-Hour-Call within the regular surgical schedule
  Other Names: LapSim

SUMMARY:
The study aimed to evaluate the effects of 24-Hour-Call-associated acute partial sleep deprivation on surgical residents' technical and cognitive performance in a virtual reality (VR) setting. Physiological parameters were used to quantify fatigue in respect to hours of sleep and subjective degrees of sleepiness. Technical performance and cognitive skills were assessed through low- and high fidelity tasks usig the VR- simulator LapSim. Objective alertness was measured by the standardized d2-Paper-Pencil-Test. Cited assessments were performed on three consecutive mornings- pre- and post-call as after 24 hours resting.

DETAILED DESCRIPTION:
Summary Background Data:

The effect of acute partial sleep deprivation on surgical proficiency is still controversially discussed. The present study is the first to measure objective physiological parameters of fatigue in respect to subjective perceptions of sleepiness in VR- research of surgical performance.

Methods:

38 surgeons were explored on three consecutive mornings: prior to a 24-Hour- Call, post-call and after 24 hours resting. Hours of sleep were recorded. Subjective alertness was assessed using the standardized Stanford-Sleepiness-Scale (SSS). Saliva cortisol concentrations and pupillary activity were measured by ELISA and pupillography. The VR-simulator LapSim® was used to assess technical skills through defined low- fidelity VR-tasks "cutting", "clip applying" and cognitive skills through defined high-fidelity VR-tasks "intracorporal suturing", "VR-cholecystectomy". Objective alertness was measured by the standardized d2-Paper-Pencil-Test.

ELIGIBILITY:
Inclusion Criteria:

* Surgical interns, junior- or senior residents
* Successful completion of a minimum of 10 basic VR- tasks with the VR- simulator LapSim: "camera navigation", "coordination", "clip applying", "Cutting", and "diathermy cutting" and a minimum of 5 sessions of advanced VR- tasks: "fine dissection", "intracorporal suturing" and "VR- cholecystectomy"
* Voluntary participation
* Written informed consent

Exclusion Criteria:

* Lack of required VR- training
* Lack of informed consent

Ages: 28 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * 38 surgeons (20 male, 18 female)
  * 4 senior registrars, 15 junior registrars, 19 interns
  * age 24-48 years; mean 30 years
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Technical and cognitive performance | 3 days
  Technical and cognitive performance was assessed in a VR-setting of defined parameters of performance and the d2-Paper-Pencil-Test on three consecutive mornings- pre- and post call and after 24 hours resting.

SECONDARY OUTCOMES:
Sleepiness and Fatigue | 4 months
  Sleepiness was assessed by Stanford Sleepiness Sclae (SSS) and fatigue was measured through pupillography and saliva cortisol concentration on three consecutive mornings- pre- and post call and after 24 hours resting.

CONTACTS AND LOCATIONS:
Overall Officials: Katja KM Maschuw, MD, Principal Investigator — Philipps University Marburg
Locations (1):
- Department of Visceral-, Thoracic- and Vascular Surgery, Univeristy Hospital Giessen and Marburg- Location Marburg, Marburg, Hesse, Germany